CLINICAL TRIAL: NCT06588413
Title: Randomized, Double-Blind Study of FOND (Fosaprepitant, ONdansetron, Dexamethasone) Plus Either Olanzapine 2.5 mg Versus 5 mg for the Prevention of Chemotherapy Induced Nausea and Vomiting in Patients Receiving High-dose Melphalan Conditioning: The FONDO-LOW Study
Brief Title: Olanzapine 2.5 vs 5 mg in Quadruplet Nausea/Vomiting Prophylaxis Before High-Dose Melphalan
Acronym: FONDO-LOW
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Amber Clemmons, Professor / Clinical Pharmacy Specialist, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2216424
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma; Autologous Stem Cell Transplantation
Keywords: CINV; Nausea; Olanzapine; Melphalan; autologous transplant
MeSH Terms: conditions — Multiple Myeloma; Nausea | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olanzapine 2.5 mg (Experimental): Olanzapine 2.5 mg dose to be given on the day of high-dose melphalan and three days after
  Interventions: Drug: Olanzapine
- Olanzapine 5 mg (Active Comparator): Olanzapine 5 mg dose to be given on the day of high-dose melphalan and three days after
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Subjects will be randomized to either olanzapine 2.5 mg or 5 mg
  Other Names: Zyprexa

SUMMARY:
Patients who receive a chemotherapy called melphalan are at high risk of having nausea and vomiting. A medication called olanzapine has been shown to decrease nausea and vomiting after chemotherapy. A previous research study found the 10 mg dose of olanzapine (combined with 3 standard medications used routinely to prevent nausea/vomiting) to be effective for patients who received melphalan chemotherapy, but several other studies have shown many patients have a side effect of sleepiness (e.g., sedation) with that dose of the medication. Our study will compare two lower doses of olanzapine (5 mg and 2.5 mg) in combination with the 3 standard medications used to prevent nausea/vomiting in the patients who receive melphalan chemotherapy to determine which dose is effective in preventing nausea and vomiting with the lowest amount of sleepiness side effect.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded trial comparing olanzapine 2.5 mg vs 5 mg in combination with standard triplet antiemetic prophylaxis in patients with multiple myeloma who are receiving high-dose melphalan conditioning chemotherapy before autologous stem cell transplantation to determine chemotherapy-induced nausea and vomiting (CINV) and sedation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of high-dose melphalan 140-200 mg/m2
* Autologous stem cell transplantation recipient

Exclusion Criteria:

* Allergy to olanzapine
* Documented nausea or vomiting within 24 hours prior to enrollment
* Treatment with other antipsychotic agents such as risperidone, quetiapine, clozapine, phenothiazine, or butyrophenone within 30 days prior to enrollment or planned during protocol therapy
* Chronic alcoholism
* Pregnant
* Decline or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Complete Response | From day of chemotherapy (acute phase) through 5 days after chemotherapy (delayed phase)
  The primary objective is to compare the percentage of patients achieving chemotherapy-induced nausea and vomiting (CINV) complete response (CR), where CR is defined as no emesis and no more than mild nausea (</=1 score on a 4-point categorical scale [0 = none, 1 = mild, 2 = moderate, and 3 = severe]) during the overall assessment period (defined as the day of chemotherapy through 5 days after chemotherapy).

SECONDARY OUTCOMES:
Complete Protection | From day of chemotherapy (acute phase) through 5 days after chemotherapy (delayed phase)
  Complete protection (CP) defined as no emesis, no more than mild nausea, and no use of breakthrough antiemetic agents
Incidence of patients with no more than minimal sedation | From day of chemotherapy (acute phase) through 5 days after chemotherapy (delayed phase)
Incidence of patients with no more than minimal nausea | From day of chemotherapy (acute phase) through 5 days after chemotherapy (delayed phase)
Number of emetic episodes | From day of chemotherapy (acute phase) through 5 days after chemotherapy (delayed phase)
Number of breakthrough antiemetic doses | From day of chemotherapy (acute phase) through 5 days after chemotherapy (delayed phase)

CONTACTS AND LOCATIONS:
Locations (1):
- Wellstar MCG, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bajpai J, Kapu V, Rath S, Kumar S, Sekar A, Patil P, Siddiqui A, Anne S, Pawar A, Srinivas S, Bhargava P, Gulia S, Noronha V, Joshi A, Prabhash K, Banavali S, Sarin R, Badwe R, Gupta S. Low-dose versus standard-dose olanzapine with triple antiemetic therapy for prevention of highly emetogenic chemotherapy-induced nausea and vomiting in patients with solid tumours: a single-centre, open-label, non-inferiority, randomised, controlled, phase 3 trial. Lancet Oncol. 2024 Feb;25(2):246-254. doi: 10.1016/S1470-2045(23)00628-9. Epub 2024 Jan 12. PMID 38224701
- [Background] Clemmons AB, Orr J, Andrick B, Gandhi A, Sportes C, DeRemer D. Randomized, Placebo-Controlled, Phase III Trial of Fosaprepitant, Ondansetron, Dexamethasone (FOND) Versus FOND Plus Olanzapine (FOND-O) for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Patients with Hematologic Malignancies Receiving Highly Emetogenic Chemotherapy and Hematopoietic Cell Transplantation Regimens: The FOND-O Trial. Biol Blood Marrow Transplant. 2018 Oct;24(10):2065-2071. doi: 10.1016/j.bbmt.2018.06.005. Epub 2018 Jun 13. PMID 29906570